CLINICAL TRIAL: NCT04273542
Title: Multicenter Large-scale Validation Study of the Interest of Broadband Spectroscopy Analysis (Femto/Attosecond by Infrared Laser) on Liquid Biopsies in Breast Cancer Screening
Brief Title: Interest of Broadband Spectroscopy Analysis by Infrared Laser on Liquid Biopsies in Breast Cancer Screening
Acronym: ICRG0101
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: International Cancer Research Group, United Arab Emirates (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A00058-31
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Female; BRCA1 Mutation; BRCA2 Mutation
Keywords: Breast cancer; broadband spectroscopy laser; liquid biospsies; cancer screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control cohort (Other): In this cohort, women recruited participated to organised breast cancer screening. They must not have an invasive breast cancer.
  They will have 3 liquid biopsy : the first at inclusion and then at each mammogram every two years (organised breast cancer screening).
  Interventions: Other: liquid biopsy
- Patient cohort (Other): In this cohort, women for who an invasive breast cancer has been diagnose will be included.
  Only one liquid biopsy will be collected before any treatment.
  Interventions: Other: liquid biopsy
- Exploratory cohort (Other): In this cohort, women with high risk of BRCA1/2 mutation but without invasive breast cancer.
  6 liquid biopsies will be collected : each year after inclusion during 5 years.
  Interventions: Other: liquid biopsy

INTERVENTIONS:
Other: liquid biopsy — Blood sample collection during follow-up of the three cohorts of patients

SUMMARY:
The purpose of this study is to validate the interest of broadband spectroscopy analysis (femto/attosecond by infrared laser) on liquid biopsies in breast cancer screening.

DETAILED DESCRIPTION:
Each patient will have one or more liquid biopsy during the follow-up according to the cohort and have a mammogram at the same time.

Biopsies will be analysed by broadband spectroscopy in order to compare the results to mammogram result.

ELIGIBILITY:
Inclusion Criteria:

*For all participants :

* Adult woman capable of giving informed consent to research participation
* Affiliation to the French social security system

  >For Control cohort:
* Woman participating in organised screening or benefiting from individual follow-up, eligible as such for a mammogram

  >For Patient cohort:
* woman with invasive breast cancer T0N1, T1N0-1, T2N0-1 (histologically proven) at inclusion and before any cancer treatment

  >For Exploratory cohort:
* woman carrying the BRCA1/2 mutation, followed according to standard recommendations or
* woman carrying the BRCA1/2 mutation suffering from in situ BC discovered on biopsy and histologically confirmed

Exclusion Criteria:

* For all participants :

  * Refusal to participate
  * Reluctant or unable to comply with study requirements
  * Pregnant or breastfeeding woman
  * History of breast cancer
* For Patient cohort

  - Patients with Stage III/IV or Bilateral Breast Cancer
* For Control cohort:

  * Invasive breast cancer suspected at mammography before liquid biopsy*
  * Mammography classified ACR3 or ACR4
* For Exploratory cohort:

  * Concomitant breast cancer

    * At inclusion visit, woman for whom an invasive breast cancer will be suspected at mammography will be include in Patient cohort after an histological proof of cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Validation of the value of molecular profiling analysis in broadband laser spectroscopy on liquid biopsies for breast cancer screening | Comparison between the different cohorts at (T0 : inclusion) and the others visits (T1:+1year; T2: +2years; T3 : +3years; T4:+4years; T5: 5years)
  To validate the value of molecular profiling analysis in broadband laser spectroscopy on liquid biopsies for invasive breast cancer screening by comparing a cohort of patients with localized invasive breast cancer (Stage I/II) to a cohort of women without invasive breast cancer from organized or individual age-matched screening.

SECONDARY OUTCOMES:
Correlating the results of high-speed laser spectroscopy analysis on liquid biopsies with mammography data (ACR 0-5) | T0: inclusion; T1:+1year; T2: +2years; T3 : +3years; T4:+4years; T5: 5years
  The results of high-speed laser spectroscopy analysis on liquid biopsies will be correlated with mammography data
Estimate detection rate of both breast cancer screening methods (spectroscopy/mammography) for control cohort | T0 : inclusion; T2 : +2 years; T4: +4years
  Estimate the rate of detection of invasive breast cancer occurring within 5 years of examination in the control group according to the reference method (mammography) and the innovative method ("n-variable molecular profiles") from the baseline analysis performed at Max Planck Institute and algorithmic analysis
To study the role of confounding factors in the structure of molecular profiles derived from broadband laser spectroscopy | T0: inclusion; T1:+1year; T2: +2years; T3 : +3years; T4:+4years; T5: 5years
  To study the confounding role of hormonal status and concomitant inflammatory states in the structure of molecular profiles derived from broadband laser spectroscopy
Comparison of BRCA1/2 patients molecular profiles with control and patient cohorts derived from broadband laser spectroscopy | T0: inclusion; T1:+1year; T2: +2years; T3 : +3years; T4:+4years; T5: 5years
  To study the molecular profiles derived from broadband laser spectroscopy on liquid biopsies in a cohort of high-risk women (BRCA1/2) not carrying invasive breast cancer, and to compare their positioning in relation to the 2 main cohorts of the study (patients carrying invasive breast cancer without mutation and controls without invasive breast cancer).

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique PENAULT-LLORCA, Pr, Principal Investigator — Centre Jean Perrin
Locations (9):
- France (9):
  - Centre Jean PERRIN, Clermont-Ferrand, Puy de Dome
  - La Chataigneraie (Selimed 63), Beaumont, Puy de Dôme
  - Pôle Santé République, Clermont-Ferrand, Puy de Dôme
  - Institut de Cancérologie de l'Ouest, Angers
  - Centre Eugène MARQUIS, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Hôpital La Pitié Salpêtrière, Paris, Île-de-France Region
  - Hôpital Saint-Louis, Paris, Île-de-France Region
  - Hôpital Tenon, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No